CLINICAL TRIAL: NCT05766163
Title: Comparative Evaluation of New Surgical Robotic Platforms for the Radical Prostatectomy Procedure
Brief Title: Comparison of Outcomes of Multiple Platforms for Assisted Robotic - Prostate
Acronym: COMPAR-P
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliera Universitaria Integrata Verona (Other)
Responsible Party: Principal Investigator, Alessandro Antonelli, MD, Prof, Director of Urology Unit, Azienda Ospedaliera Universitaria Integrata Verona
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: COMPAR-P
Record Dates: First submitted 2023-02-13; First posted 2023-03-13 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Prostate Cancer
Keywords: Robotic-assisted surgery; Prostatectomy; Multiple surgical platforms; Postoperative complications; Operative outcomes
MeSH Terms: conditions — Prostatic Neoplasms; Postoperative Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- DaVinci system (Active Comparator): Robot-assisted radical prostatectomy is carried out through daVinci platform.
  Interventions: Device: DaVinci RARP
- Hugo system (Experimental): Robot-assisted radical prostatectomy is carried out through Hugo platform.
  Interventions: Device: Hugo RARP
- Versius system (Experimental): Robot-assisted radical prostatectomy is carried out through Versius platform.
  Interventions: Device: Versius RARP

INTERVENTIONS:
Device: DaVinci RARP — Assisted-robotic radical prostatectomy.
  Other Names: DaVinci® Surgical System
  Arms: DaVinci system
Device: Hugo RARP — Assisted-robotic radical prostatectomy.
  Other Names: Hugo™ RAS System
  Arms: Hugo system
Device: Versius RARP — Assisted-robotic radical prostatectomy.
  Other Names: Versius® Robotic Surgery System
  Arms: Versius system

SUMMARY:
The object of this exploratory clinical trial is to evaluate post-operative complications in a population that underwent Robotic Assisted Radical Prostatectomy (RARP) made with multiple platforms:

* DaVinci;
* Hugo;
* Versius.

The questions it aims to answer are:

* Does the estimation of the post-operative complications suggest something?
* Are differences (intra-operative, post-operative, oncological, functional, technical, and economic) among the three intervention approaches observable?

Participants will be invited to fill out questionnaires and join one of these three groups:

1. surgery with the daVinci platform;
2. surgery with the Hugo platform;
3. surgery with the Versius platform.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 and < 90 years;
* Organ-localized prostate cancer with a surgical indication of radical prostatectomy;
* Informed consent provided.

Exclusion Criteria:

* Age < 18 and > 90 years;
* Contraindication to radical prostatectomy procedure;
* Non-organ confined prostate cancer;
* Refusal to participate.

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-03-14 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Number of participants with postoperative complications | Over the 4 days post surgery
  Overall postoperative complications (% score >0) are considered by Clavien-Dindo Classification 7 grades (I, II, IIIa, IIIb, IVa, IVb and V): the higher the grade, the higher the severity of the complication
Number of participants with moderate to major postoperative complications | Over the 4 days post surgery
  Moderate to major complications (% score >=2) are considered by Clavien-Dindo Classification 7 grades (I, II, IIIa, IIIb, IVa, IVb and V): the higher the grade, the higher the severity of the complication
Number of participants with major postoperative complications | Over the 4 days post surgery
  Major complications (% score >=3) are considered by Clavien-Dindo Classification 7 grades (I, II, IIIa, IIIb, IVa, IVb and V): the higher the grade, the higher the severity of the complication

SECONDARY OUTCOMES:
Estimated Blood Loss | Intraoperative
  Volume
Overall duration of the surgery | Intraoperative
  Minutes
Anesthesia, Lymphadenectomy, Prostatectomy | Entrance of patient into operating room until completion of surgery
  Minutes
Number and type of intraoperative complications | Intraoperative
  Note
Postoperative hospitalization | From the surgery day up to 10 days postoperative
  Days of recovery until the date of release
Postoperative pain | 1-4 days postoperative
  Numerical Rating Scale (NRS) 0-10 scale for the self-reported rate of pain: zero meaning "no pain" and 10 meaning "the worst pain imaginable"
Prostate Specific Antigen (PSA) | 1 month follow-up
  PSA test
Positive Surgical Margin | Up to 2 weeks postoperative (during histological analysis)
  Rate at histological examination
Lymph nodes resection | Intraoperative
  Number of lymph nodes removed
Urinary, sexual, and intestinal function assessment | Preoperative and follow-up (1, 3 and 6 months)
  University of California, Los Angeles (UCLA) Prostate Cancer Index (PCI) questionnaire
  Domains:
  * Urinary function (5 items)
  * Urinary bother (1 item)
  * Sexual function (8 items)
  * Sexual bother (1 item)
  * Bowel function (4 items)
  * Bowel bother (1 item)
  Response options: 3- to 6-point Likert scales. The higher the score, the better the outcome
Quality of Life Evaluation | Preoperative and follow-up at 1, 3 and 6 months
  Short Form Health Survey (SF-36) 36 questions (8 domains) for self-reported measure of health. Domain score from 0 to 100: the higher the score, the more favorable the state of health
Time taken for platform-related technical steps | From the room setting, through surgical procedure until postoperative room restoration for each of expected 150 surgeries (through study completion: an average of 1 year)
  Set up of operating table, Electric connections, Draping, Undraping, Docking, Undocking, Cleaning: time in minutes
Possible malfunction of the platform | Intraoperative
  Note
Procedure-related costs | From surgical procedure to the end of follow-up period (6 months)
  Estimate

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro AA Antonelli, Principal Investigator — Azienda Ospedaliera Universitaria Integrata Verona
Locations (1):
- Urology Unit, AOUI Verona, Verona, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/35156838/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/32169362/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/35047788/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/29442240/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/33559802/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/16846677/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/21427584/